CLINICAL TRIAL: NCT02031068
Title: Active Rehabilitation for Slow to Recover Adolescents Following Sport-Related Concussion: A Randomized Control Trial
Brief Title: Exercise for Adolescents Following Sport-Related Concussion: A Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H12-01780
Record Dates: First submitted 2013-12-10; First posted 2014-01-09 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Sport-related Concussion; Concussion; Mild Traumatic Brain Injury (MTBI)
Keywords: active rehabilitation; exercise; concussion
MeSH Terms: conditions — Brain Concussion; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Treatment-as-usual (TAU) (Active Comparator): The TAU program will be implemented after the initial assessment. It will consist of 2 components:
  1. An initial education session by an occupational therapist, relating to outcome from concussion and managing symptoms
  2. A school consultation to provide teacher education, recommend accommodations, and facilitate return to school
  Interventions: Behavioral: Treatment-as-usual (TAU)
- Behavioral:Active Rehabilitation Program (Experimental): The active rehabilitation program will be implemented for a maximum of 6-8 weeks. Each participant will be followed by regular weekly telephone calls or personal follow-up relating to outcome from concussion and managing symptoms. The participant will receive TAU (above) in addition to the 4 components listed below:
  1. Sub-maximal aerobic training for up to 15 minutes
  2. Light coordination and sport-specific exercises for up to 10 minutes
  3. Visualization and imagery techniques
  4. Home program.
  A physiotherapist will supervise the rehabilitation.
  Interventions: Behavioral: Active Rehabilitation Program

INTERVENTIONS:
Behavioral: Active Rehabilitation Program — The active rehabilitation program will be implemented for a maximum of 6-8 weeks. Each participant will be followed by regular weekly telephone calls or personal follow-up relating to outcome from concussion and managing symptoms. The participant will receive TAU (above) in addition to the 4 components listed below:
  1. Sub-maximal aerobic training for up to 15 minutes
  2. Light coordination and sport-specific exercises for up to 10 minutes
  3. Visualization and imagery techniques
  4. Home program
  A physiotherapist will supervise the rehabilitation.
  Arms: Behavioral:Active Rehabilitation Program
Behavioral: Treatment-as-usual (TAU) — The TAU program will be implemented after the initial assessment. It will consist of 2 components:
  An initial education session by an occupational therapist, relating to outcome from concussion and managing symptoms A school consultation to provide teacher education, recommend accommodations, and facilitate return to school
  Arms: Treatment-as-usual (TAU)

SUMMARY:
To test the safety and feasibility of a new treatment for adolescents who are slow to recover from a sport-related concussion, the investigators are conducting a randomised controlled trial comparing treatment as usual with an active rehabilitation program that involves sub-symptom threshold cardiac exertion, sport-specific coordination activities, and positive visualisation techniques.

DETAILED DESCRIPTION:
Most adolescents recover within the first month following a sport-related concussion. However, some do not. Little is known about how to best facilitate recovery when symptoms do not resolve spontaneously and swiftly. Although active rehabilitation has been recently suggested as a promising means of promoting recovery, current literature does not provide adequate evidence for safe adaptation into clinical practice.

Objective: The purpose of this project is to evaluate an active rehabilitation protocol for adolescents who are slow to recover following sport-related concussion. Primary aims: to confirm the tolerability and safety of the active rehabilitation protocol as compared to treatment as usual controls. Secondary aims: 1) to document the impact of active rehabilitation on post-concussion symptoms and return to activity; 2) to explore the intervention effects on quality of life, mood, energy level, balance, cognitive functioning, and return to pre-injury activities.

Study design: A parallel group open label randomized comparison trial of 30 adolescents who are slow to recover following sport-related concussion. After initial screening and assessment, both groups will receive treatment as usual. Participants in the experimental group will also participate in sub-symptom threshold exercise, sport-specific coordination practice, and positive visualisation daily.

Outcome measures: The investigators will monitor for adverse events and assess post-concussion symptoms throughout the study as a primary marker of recovery. The investigators will also report secondary outcomes such as quality of life, mood, energy level, balance and cognitive functioning. Finally the investigators will record rates of return to school (full time, part time) and rates of return to sport (regular pre-injury vs. modified level). As a result, clinicians will be able to follow a new rehabilitation protocol in a safe and meaningful way. Lastly, research findings will be disseminated in the form of a publication, at conferences, and via in-services.

Hypotheses:

1a. The drop-out rate will be comparable in the groups receiving treatment-as-usual (TAU) only versus TAU plus active rehabilitation.

1b. Adverse events occurring outside of the clinic will be comparable in the groups receiving TAU only versus TAU plus active rehabilitation.

1c. For the group receiving active rehabilitation, symptom exacerbations in the in-clinic exercise sessions will resolve within 30 minutes.

2. Participants receiving active rehabilitation will report greater improvement of post-concussion symptoms (primary outcome) at follow-up.

3. Participants receiving active rehabilitation will report higher quality of life, fewer depressive symptoms, and higher energy levels; demonstrate better balance and neuropsychological performance at follow-up; and return to their pre-injury activities at higher rates.

ELIGIBILITY:
Adolescents referred to G. F. Strong Rehabilitation Centre (GFS) for atypical recovery preventing them from entering standard return to activities protocols will be recruited on a voluntary basis to participate in this study.

Eligibility criteria for study entry are as follows:

1. sustained an injury in sports,
2. are 4 weeks post injury,
3. report 2+ persistent post-concussion symptoms with no significant improvement over the past week,
4. are between the ages of 14 and 18,
5. have no developmental, congenital, or cognitive diagnoses,
6. have no active mental health disorders,
7. are able to attend at GFS,
8. speak English as their dominant language,
9. have no prior moderate or severe TBI,
10. have no concussion in the 6 months before the present injury, and
11. medical clearance by the study physician.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Symptom Report | Baseline
  The Post-Concussion Scale consists of 22 subjectively-experienced symptoms (e.g., headache, dizziness, concentration problems, and fogginess). A total score is derived from this 22-item scale. Athletes report symptoms based on the severity of each symptom that day, allowing tracking of symptoms over very short intervals
Symptom Report | At 8 weeks (end-of-treatment)

SECONDARY OUTCOMES:
Mood | Baseline
  The Beck Depression Inventory for Youth-Second Edition is a 20-item depression screening test designed for children and adolescents.
Energy level | Baseline
  Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale will be used to monitor fatigue in the study participants, another commonly reported complaint after a MTBI. The PedsQL was designed to measure fatigue in pediatric patients; it includes a General Fatigue Scale (6 items), Sleep/Rest Fatigue Scale (6 items), and Cognitive Fatigue Scale (6 items).
Balance Testing | Baseline
  The Balance Error Scoring System (BESS) is a commonly used measure of static balance and postural stability. The test is rapid, relatively easy-to-administer, and inexpensive. A combination of three stances (narrow double leg stance; single leg stance; and tandem stance) and footing surfaces (firm surface/floor or medium density foam) are used for the test. Each stance is held, with hands on hips and eyes closed, for 20 seconds. "Error" points are given for specific behaviors, including opening eyes, lifting hands off hips, or stepping, stumbling, or falling.
  Safety Issue: Falls and fall-related injuries. Testing will be supervised by a registered physiotherapist.
Neurocognitive Testing | Baseline
  ImPACT is a computerized neuropsychological test battery that consists of six individual test modules that measure multiple aspects of cognitive functioning including attention, memory, working memory, visual scanning, reaction time, and processing speed. The test takes 20-25 minutes. Four composite (i.e., summary) scores are tabulated based upon these individual test scores: Verbal Memory, Visual Memory, Reaction Time, and Processing Speed.
Return to School and Sport | Baseline
  Number of days away from school and sports will be documented. School status will also be rated as part-time, full-time, and with/without accommodations at different time intervals.
Mood | At 8 weeks (end-of-treatment)
  The Beck Depression Inventory for Youth-Second Edition will be used
Energy level | At 8 weeks (end-of-treatment)
  Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale will be used
Balance Testing | At 8 weeks (end-of-treatment)
  The Balance Error Scoring System (BESS) will be used
Neurocognitive Testing | At 8 weeks (end-of-treatment)
  ImPACT will be used.
Return to School and Sport | At 8 weeks (end-of-treatment)
  Number of days away from school and sports will be documented. School status will also be rated as part-time, full-time, and with/without accommodations at different time intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chan, Physiotherapy, Principal Investigator — GF Strong Rehab Centre - Vancouver Coastal Health Research Institute; Grant Iverson, Ph.D, Principal Investigator — University of British Columbia, Department of Psychiatry
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Chan C, Iverson GL, Purtzki J, Wong K, Kwan V, Gagnon I, Silverberg ND. Safety of Active Rehabilitation for Persistent Symptoms After Pediatric Sport-Related Concussion: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):242-249. doi: 10.1016/j.apmr.2017.09.108. Epub 2017 Oct 5. PMID 28989074